CLINICAL TRIAL: NCT07210242
Title: Clinical Study on Monitoring Cytomegalovirus (HCMV) Reactivation After Allogeneic Hematopoietic Stem Cell Transplantation Using High-Performance miRNA Quantification Technology (PSTM-qPCR)
Brief Title: HCMV-miRNA Monitoring After Allogeneic Hematopoietic Stem Cell Transplantation Using PSTM-qPCR
Acronym: HSCT-HCMV01
Status: Not yet recruiting | Type: Observational
Sponsor: Ting YANG (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Xiamen University (Other)
Responsible Party: Sponsor-Investigator, Ting YANG, Chief Physician, Department of Hematology, Fujian Medical University First Affiliated Hospital, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: HSCT-HCMV01; FJMU(2025)648 (Other: Fujian Medical University First Affiliated Hospital)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus Infections; Hematopoietic Stem Cell Transplantation; Virus Reactivation; Graft vs Host Disease
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; Human Cytomegalovirus; MicroRNA; HCMV-miRNA; PSTM-qPCR; Viral Reactivation; Infection Monitoring; Early Diagnosis; Biomarker; GVHD
MeSH Terms: conditions — Cytomegalovirus Infections; Graft vs Host Disease; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Peripheral blood samples (10 mL EDTA-anticoagulated) will be collected from both HSCT recipients and their donors. Whole blood and separated plasma will be retained for HCMV-miRNA and HCMV-DNA testing. In addition, residual hematopoietic stem cell samples from donors will be preserved. All samples will be stored at -20°C or below and shipped on dry ice to the central laboratory at Xiamen University (National Institute of Diagnostics and Vaccine Development in Infectious Diseases) for unified testing and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allo-HSCT Recipients and Donors: Participants are patients scheduled to undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT), with stem cell sources including peripheral blood stem cells and/or bone marrow plus peripheral blood. All participants must voluntarily join the study, be able to understand study procedures, and provide written informed consent.
  This is an observational cohort with no experimental intervention. Participants will receive standard of care treatment for allo-HSCT. Blood samples (whole blood and plasma) will be collected before conditioning, during transplantation, and regularly after transplantation (weekly in months 1-3, monthly in months 4-6, and as clinically indicated up to 12 months). HCMV-miRNA and HCMV-DNA will be tested using PSTM-qPCR and conventional qPCR, respectively. Clinical outcomes such as HCMV infection/reactivation, GVHD, survival, and infection-related complications will be monitored.

SUMMARY:
Human cytomegalovirus (HCMV) infection is one of the most common and serious complications after allogeneic hematopoietic stem cell transplantation (allo-HSCT). Standard monitoring uses HCMV DNA testing, but this method may not detect the virus early enough to guide timely treatment.

This multicenter observational study will evaluate a new high-performance microRNA (miRNA) detection technology (PSTM-qPCR) for monitoring HCMV infection in allo-HSCT patients. Approximately 300 patients and their donors will be enrolled across several major transplant centers in China. Blood samples will be collected before and after transplantation to test for both HCMV-miRNA and HCMV-DNA. The study will compare the sensitivity and timing of miRNA detection with conventional DNA testing and explore whether miRNA can serve as an early biomarker of infection and related complications.

The goal is to improve early diagnosis and management of HCMV infection, reduce infection-related complications, and ultimately improve survival outcomes in patients undergoing allo-HSCT.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potentially curative treatment for hematologic malignancies and non-malignant disorders. However, post-transplant immune suppression and delayed immune reconstitution make patients highly susceptible to opportunistic infections, among which human cytomegalovirus (HCMV) infection and reactivation are the most frequent and clinically significant. HCMV reactivation has been associated with increased non-relapse mortality, graft-versus-host disease (GVHD), marrow suppression, and organ-specific disease, significantly affecting patient outcomes.

Current standard monitoring relies on quantitative polymerase chain reaction (qPCR)-based HCMV DNA testing in peripheral blood. While this method has improved patient management, limitations remain. HCMV DNA testing may lack sufficient sensitivity to detect early viral reactivation, leading to missed opportunities for timely pre-emptive therapy. Increasing evidence suggests that HCMV-encoded microRNAs (miRNAs), which play critical roles in viral latency, replication, and immune evasion, may serve as novel biomarkers for earlier detection of HCMV activity.

This prospective, multicenter, observational cohort study will evaluate the diagnostic and predictive performance of HCMV-miRNAs using a novel high-performance detection platform, PSTM-qPCR, developed in collaboration with the National Institute of Diagnostics and Vaccine Development in Infectious Diseases at Xiamen University. PSTM-qPCR offers markedly improved sensitivity and specificity compared with conventional qPCR, with the ability to distinguish single-base differences and detect viral activity earlier.

Approximately 300 allo-HSCT recipients and their donors will be enrolled across seven transplant centers in China. Blood samples will be collected at baseline (pre-transplant) and serially post-transplant (weekly during the first 3 months, monthly through 6 months, and as clinically indicated up to 12 months). Both HCMV-miRNA and HCMV-DNA will be measured. Primary outcome measures include the diagnostic performance of HCMV-miRNA compared with HCMV-DNA for early detection of HCMV infection. Secondary outcomes include rates of HCMV infection and reactivation, HCMV-related mortality and organ disease, GVHD incidence, and overall survival.

The study aims to validate HCMV-miRNA as a reliable early biomarker for HCMV infection in allo-HSCT recipients. By establishing a sensitive and clinically applicable monitoring strategy, this research seeks to improve infection control, guide individualized antiviral therapy, and ultimately enhance survival and quality of life in transplant patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled to undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT).

Stem cell source includes peripheral blood stem cells and/or bone marrow plus peripheral blood.

Ability to understand study procedures and provide written informed consent.

Voluntary participation in the study.

Exclusion Criteria:

* Pregnant or breastfeeding women.

Children or individuals with severe cognitive impairment who cannot comply with blood sample collection.

Patients with severe comorbidities or other medical conditions judged by the investigator to significantly interfere with study participation or follow-up.

Withdrawal of informed consent during the study.

Clinical background or history that may introduce significant confounding effects, or when additional sampling frequency is deemed to pose undue risk to the participant.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients scheduled to undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT) at participating transplant centers in China, along with their corresponding stem cell donors. Eligible recipients are patients with hematologic malignancies or related disorders who meet transplant indications. Stem cell sources include peripheral blood stem cells and/or bone marrow plus peripheral blood. All participants must voluntarily join the study and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2028-10-10 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of HCMV-miRNA compared with HCMV-DNA | From pre-conditioning (baseline, before allo-HSCT) through 12 months post-transplantation
  Evaluate the diagnostic accuracy of HCMV-miRNA detection (using PSTM-qPCR) compared with conventional HCMV-DNA testing for early identification of cytomegalovirus infection or reactivation in allo-HSCT recipients. Outcome measures include sensitivity, specificity, and time to first positive result.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and ethical restrictions. Only de-identified, aggregated results will be published in scientific journals or presented at academic conferences.

REFERENCES:
- [Background] Toyooka S, Ito M, Kakinuma A, Kayama S, Watanabe K, Miyamoto W, Nakagawa T, Kawano H. Periarticular multimodal drug injection does not improves early postoperative analgesia compared with continuous interscalene brachial plexus block after arthroscopic rotator cuff repair: A retrospective single-center comparative study. J Orthop Sci. 2020 May;25(3):405-409. doi: 10.1016/j.jos.2019.04.013. Epub 2019 May 29. PMID 31153741
- [Background] Pujari A, Kumar S, Markan A, Chawla R, Damodaran S, Kumar A. Buckling surgery on a goat's eye: A simple technique to enhance residents' surgical skill. Indian J Ophthalmol. 2019 Aug;67(8):1327-1328. doi: 10.4103/ijo.IJO_1779_18. PMID 31332123
- [Background] Lyons MS, Kunnathur VA, Rouster SD, Hart KW, Sperling MI, Fichtenbaum CJ, Sherman KE. Prevalence of Diagnosed and Undiagnosed Hepatitis C in a Midwestern Urban Emergency Department. Clin Infect Dis. 2016 May 1;62(9):1066-71. doi: 10.1093/cid/ciw073. Epub 2016 Feb 21. PMID 26908799
- [Background] Li L, Liu Y, Chen Y, Zhai W, Dai Z. Research progress on layered metal oxide electrocatalysts for an efficient oxygen evolution reaction. Dalton Trans. 2024 May 28;53(21):8872-8886. doi: 10.1039/d4dt00619d. PMID 38738345
- [Background] Melnik S, Gabler J, Dreher SI, Hecht N, Hofmann N, Grossner T, Richter W. MiR-218 affects hypertrophic differentiation of human mesenchymal stromal cells during chondrogenesis via targeting RUNX2, MEF2C, and COL10A1. Stem Cell Res Ther. 2020 Dec 10;11(1):532. doi: 10.1186/s13287-020-02026-6. PMID 33303006
- See also: National Institute of Diagnostics and Vaccine Development in Infectious Diseases, Xiamen University (Collaborator, central laboratory for HCMV-miRNA testing). — https://nidvd.xmu.edu.cn/
- See also: European Conference on Infections in Leukaemia (ECIL) official site, providing international guidelines on CMV management in HSCT. — https://www.ecil-leukaemia.com/
- See also: Chinese expert consensus on cytomegalovirus infection management in allogeneic HSCT (2022 edition, open access). — https://pmc.ncbi.nlm.nih.gov/articles/PMC9593016/